CLINICAL TRIAL: NCT03604835
Title: Mucopolysaccharidosis VII Disease Monitoring Program (MPS VII DMP)
Brief Title: Mucopolysaccharidosis VII Disease Monitoring Program
Status: Recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX003-CL401; EUPAS25082 (Other: EU PAS Number)
Record Dates: First submitted 2018-07-18; First posted 2018-07-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis VII; MPS VII; MPS 7; Sly Syndrome
Keywords: UX003; Mepsevii; vestronidase alfa-vjbk; vestronidase alfa; recombinant human beta-glucuronidase
MeSH Terms: conditions — Mucopolysaccharidosis VII

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MPS VII receiving vestronidase-alfa: via prescription, or early access/ compassionate use program
  Interventions: Other: No Intervention
- Patients with MPS VII not receiving vestronidase-alfa: no treatment or treatment other than vestronidase alfa
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Access to any treatment is through authorized commercial use or available expanded access programs only and not as a part of this DMP.

SUMMARY:
The objectives of this study are to characterize MPS VII disease presentation and progression and assess long-term effectiveness and safety, including hypersensitivity reactions and immunogenicity of vestronidase alfa.

DETAILED DESCRIPTION:
The Mucopolysaccharidosis VII Disease Monitoring Program (MPS VII DMP) is a global, prospective, multicenter, longitudinal protocol designed to characterize MPS VII disease presentation and progression, assess long-term effectiveness and safety of vestronidase alfa, including hypersensitivity reactions and immunogenicity , as well as prospectively investigate longitudinal change across biomarker(s), clinical assessments, and patient/ caregiver-reported outcome measures in a representative population. The aim of this DMP is to collect data on patients with MPS VII to provide a comprehensive dataset on the clinical presentation, heterogeneity, and disease progression, and meaningful standardized ICH GCP-quality data collected in-clinic across multiple sites globally. The DMP is not a randomized study and both treated and untreated patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPS VII based on laboratory diagnosis, including either enzymatic or mutation analysis.
* Willing and able to provide written informed consent or, in the case of patients under the age of 18 (or below adult ages as defined by local laws and regulations) or patients >18 years of age who have cognitive deficiencies, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the DMP has been explained, and prior to any research-related procedures.
* Willing to comply with DMP visit schedule.

Exclusion Criteria:

* Concurrent participation in other pharmaceutical company-sponsored interventional clinical trial unless approved by Ultragenyx.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of MPS VII, including patients who already received vestronidase alfa in an Ultragenyx clinical trial or early access/ compassionate use program, and patients not receiving vestronidase alfa.
  Patients who were previously enrolled in an Ultragenyx-sponsored clinical trial may participate in the DMP if they have completed or discontinued from the clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Course of MPS VII Disease | 10 years
  To characterize MPS VII disease presentation and progression over time in patients treated and not treated with vestronidase alfa
Long-term Effectiveness of Vestronidase Alfa | 10 years
  To evaluate longitudinal change in biomarker(s), clinical assessments and patient/caregiver reported outcomes to examine the effectiveness of vestronidase alfa
Long-term Safety of Vestronidase Alfa | 10 years
  Hypersensitivity reactions, immunogenicity and other safety outcomes will be assessed to examine the long-term safety of vestronidase alfa.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc.
Locations (14):
- United States (7):
  - Children's Hospital of Orange County, Orange, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - New York University Langone Medical Center, New York, New York
  - University of Utah Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Laboratorio de Neuroquimica Dr. N.A. Chamoles S.R.L., Buenos Aires, Buenos Aires, Argentina
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Centre Hospitalier Universitaire La Timone, Marseille, Provence-Alpes-Côte d'Azur Region, France
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Germany
- Erasmus University Medical Center Rotterdam, Rotterdam, South Holland, Netherlands
- Centro Hospitalar do Porto, Porto, Portugal
- Hospital Universitario Virgen del Rocío Pabellón Infantil, Seville, Sevilla, Spain

REFERENCES:
- See also: Ultragenyx Patient Advocacy/MPS 7 Disease Information — https://ultrarareadvocacy.com/conditions-we-study/mucopolysaccharidosis-type-vii-mps-vii/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/